CLINICAL TRIAL: NCT04608188
Title: An Intervention to Prevent Weight Gain and Unhealthy Behaviors in Children From Economically Disadvantaged Circumstances
Brief Title: Preventing Weight Gain and Unhealthy Behaviors in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, R. Glenn Weaver, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00091526
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Summer Program (Experimental): Children in the intervention will attend a summer day camp operated at their school.
  Interventions: Behavioral: Summer Camp
- No Program (No Intervention): The control children will not receive an intervention of any kind and will be asked to go about their summer as they typically would.

INTERVENTIONS:
Behavioral: Summer Camp — The intervention camps will operate according to routine practice, with no assistance from the investigative team. The camps provide indoor and outdoor opportunities for children to be physically active each day, provide enrichment and academic programming, as well as provide breakfast, lunch, and snacks. All camp meals will adhere to the United States Department of Agriculture Summer Food Service Program nutrition guidelines. The camps employ 1 staff member for every 12 children - which is consistent with childcare regulations in the state of operation and operate daily (Mon-Fri) for 8 weeks during the summer. The camps open at 7am and close 6 pm daily.
  Arms: Summer Program

SUMMARY:
This study will address engagement in unhealthy behaviors, low levels of self-regulation, and unhealthy weight gain for children from low-income households.

DETAILED DESCRIPTION:
Evidence suggests that components within structured days (e.g., school days) have a positive influence on children's obesogenic behaviors (i.e., diet, sleep, physical activity, sedentary behaviors) and self-regulation. In this pilot study children will be randomized to two arms: attend a structured summer camp, not attend a camp. The investigators hypothesize that children attending the summer camp will engage in more healthy obesogenic behaviors, display higher levels of self-regulation, and subsequently will experience less weight gain than children not attending the summer camp. To test this hypothesis the following specific aims will be accomplished: Aim 1 (Primary): Compare changes in BMI z-scores and fitness among children from low-income households attending a structured summer day camp and those not attending a structured summer day camp. Aim 2 (Secondary): Compare changes in obesogenic behaviors among children attending a structured summer day camp and those not attending a structured summer day camp. Aim 3 (Exploratory): Explore changes in self-regulation and the moderating effect of these changes on primary and secondary outcomes among children attending and not attending a structured summer day camp.

ELIGIBILITY:
Inclusion Criteria:

* participants will be boys and girls that attend one of the participating schools
* indicates "yes' on an informed consent document for participation in the study

Exclusion Criteria:

* diagnosis of an intellectual disability, such as Down Syndrome, Fragile X, Fetal Alcohol and/or a physical disability, such as wheelchair use, that prevents the ability to ambulate without assistance.
* children who plan to enroll in a summer camp during the year that they participate in the study will also be excluded from the study.
* No other exclusion criteria will be used.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weaver RG, Armstrong B, Adams E, Beets MW, White J, Flory K, Wilson D, McLain A, Tennie B. Feasibility and preliminary efficacy of structured programming and a parent intervention to mitigate accelerated summer BMI gain: a pilot study. Pilot Feasibility Stud. 2023 May 15;9(1):83. doi: 10.1186/s40814-023-01312-3. PMID 37189190
- [Derived] Weaver RG, Armstrong B, Adams E, Beets M, White J, Flory K, Wilson D, Mclain A, Tennie B. Feasibility & Preliminary Efficacy of Structured Programming and a Parent Intervention to Mitigate Accelerated Summer BMI Gain: A pilot study. Res Sq [Preprint]. 2022 Mar 29:rs.3.rs-1466063. doi: 10.21203/rs.3.rs-1466063/v1. PMID 35378750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Summer Program | No Program
Started | 21 | 68
Completed | 17 | 60
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Summer Program | No Program | Total
Number analyzed (Participants) | 21 | 68 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.5 (1.7) | 8.4 (1.4) | 8.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 30 | 41
  Male | 10 | 38 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 37 | 49
  White | 9 | 31 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 68 | 89
BMI z-score [Mean (Standard Deviation); unit: z-score] — Centers for Disease Control age and sex-specific Body Mass Index z-scores A z-score of 0 represents the population mean Higher or lower z-scores could represent better or worse outcomes as too low could be underweight and too high could indicate overweight or obesity.
  Children above the 85th percentile are considered overweight while children above the 95th percentile are considered obese
  z-score | 0.61 (1.28) | 0.91 (1.36) | 0.84 (1.33)
Inhibit BRIEF Subscale [Mean (Standard Deviation); unit: t-score] — The Behavior Rating Inventory of Executive Function was developed to provide a window into the everyday behavior associated with specific domains of the executive functions. This can be described as the ability to resist impulses and the ability to stop one's own behavior at the appropriate time. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
  t-score | 55.8 (16) | 53.7 (11.9) | 54.3 (12.9)
Monitor BRIEF Subscale [Mean (Standard Deviation); unit: t-score] — The Behavior Rating Inventory of Executive Function measures Task-oriented monitoring or work-checking habits and Self-monitoring or interpersonal awareness. The task monitoring portion of the scale captures whether a child assesses his or her own performance during tasks to ensure accuracy. The self-monitoring portion of the scale evaluates whether a child keeps track of the effect that his or her behavior has on others. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
  t-score | 53.6 (13.8) | 52.7 (11.3) | 52.9 (11.9)
Emotional Control BRIEF Subscale [Mean (Standard Deviation); unit: t-score] — The Behavior Rating Inventory of Executive Function measures The Emotional Control scale measures the impact of executive function problems on emotional expression and assesses a child's ability to modulate or control his or her emotional responses. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
  t-score | 56.8 (17.1) | 55.0 (14.1) | 55.4 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index Z-score
Description: Measure Description: Centers for Disease Control age and sex-specific Body Mass Index z-scores. A z-score of 0 represents the population mean. Higher or lower z-scores could represent better or worse outcomes as too low could be underweight and too high could indicate overweight or obesity.
  Children above the 85th percentile are considered overweight while children above the 95th percentile are considered obese
Time Frame: End of school year (start of summer - baseline), beginning of the following school year (3 month)
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Summer Program | No Program
Number analyzed (Participants) | 21 | 68
z-score | 0.04 (0.572466) | -0.14 (0.09)
Statistical Analysis 1: Comparison: No Program; Test type: Superiority; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in Inhibit BRIEF Subscale
Description: The Behavior Rating Inventory of Executive Function was developed to provide a window into the everyday behavior associated with specific domains of the executive functions. This can be described as the ability to resist impulses and the ability to stop one's own behavior at the appropriate time. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
Time Frame: End of school year (start of summer - baseline), beginning of the following school year (3 month)
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Summer Program | No Program
Number analyzed (Participants) | 21 | 68
t-score | 6.0 (5.8) | 2.3 (5.6)
Statistical Analysis 1: Comparison: No Program; Test type: Superiority; p = 0.05, Mixed Models Analysis

3. Secondary Outcome: Change in Monitor BRIEF Subscale
Description: The Behavior Rating Inventory of Executive Function measures Task-oriented monitoring or work-checking habits and Self-monitoring or interpersonal awareness. The task monitoring portion of the scale captures whether a child assesses his or her own performance during tasks to ensure accuracy. The self-monitoring portion of the scale evaluates whether a child keeps track of the effect that his or her behavior has on others. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
Time Frame: End of school year (start of summer - baseline), beginning of the following school year (3 month)
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Summer Program | No Program
Number analyzed (Participants) | 21 | 68
t-score | 8.6 (5.5) | 6.6 (6.0)
Statistical Analysis 1: Comparison: No Program; Test type: Superiority; p = 0.05, Mixed Models Analysis

4. Secondary Outcome: Change in Emotional Control BRIEF Subscale
Description: The Behavior Rating Inventory of Executive Function measures The Emotional Control scale measures the impact of executive function problems on emotional expression and assesses a child's ability to modulate or control his or her emotional responses. For T-score values 50 indicates the population mean with a standard deviation of 10 higher scores represent a worse outcome.
Time Frame: End of school year (start of summer - baseline), beginning of the following school year (3 month)
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Summer Program | No Program
Number analyzed (Participants) | 21 | 68
t-score | -0.44 (6.9) | 0.36 (7.3)
Statistical Analysis 1: Comparison: No Program; Test type: Superiority; p = 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Data were collected for the 1 year that the participants were enrolled in the study.
Description: The participants were healthy children
Arm/Group | Summer Program | No Program
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/68
Other Adverse Events (participants affected / at risk) | 0/21 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04608188/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04608188/SAP_001.pdf
  • Informed Consent Form (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04608188/ICF_002.pdf